CLINICAL TRIAL: NCT02832752
Title: The BC Extracorporeal Cardiopulmonary Resuscitation Trial for Refractory Out-of-Hospital Cardiac Arrest
Brief Title: BC ECPR Trial for Out-of-Hospital Cardiac Arrest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in Hospital Protocols and COVID-19
Sponsor: University of British Columbia (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); Physio-Control (Industry); Providence Healthcare (Other)
Responsible Party: Principal Investigator, Brian Grunau, Assistant Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H15-01701
Record Dates: First submitted 2016-06-28; First posted 2016-07-14 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECPR Region (Active Comparator): The ECPR region has incorporated ECPR therapy into the out-of-hospital cardiac arrest algorithm. Within the ECPR Protocol, full standard advanced cardiac life support treatments will continue up until the time of ECMO initiation. The anticipated enrolment in this group is 70 patients. All eligible patients in the region will be enrolled, regardless of whether the ECPR protocol is activated or whether the patient is actually treated with ECPR.
  Interventions: Procedure: ECPR Protocol
- Control Region (No Intervention): The control region will continue usual care as per current protocols which include standard advanced cardiac life support. Patients will be enrolled in the control region group at the same juncture of study eligibility. The anticipated enrolment in this group is 350 patients.
  Within BCEHS practice, transport to hospital without prior return of spontaneous circulation is rare. Termination of resuscitation must be approved by an on-call physician and cannot occur prior to 30 minutes of resuscitation efforts.

INTERVENTIONS:
Procedure: ECPR Protocol — The regional protocol is activated for eligible patients who remain pulseless after 3 cycles of resuscitation, and intubation. The hospital team is activated at this time, which includes the emergency department team, a perfusionist, and a cardiovascular surgeon. A mechanical CPR device (Lucas chest compression device) is applied at this time and the patient is transported to hospital. The goal times from first professional CPR to ECMO flows is < 60 minutes, and from emergency department (ED) arrival to ECMO flows < 30 minutes.
  Arms: ECPR Region

SUMMARY:
The addition of an Extracorporeal-Cardiopulmonary Resuscitation (ECPR) service to a region may improve the survival of young patients with sudden unexpected cardiac arrest.The primary aim of this study is to determine the benefit of the systematic integration of ECPR services into the out-of-hospital cardiac arrest management algorithm. The investigators will compare the outcomes of ECPR-eligible patients in the intervention region, in comparison to patients meeting the same criteria in a comparable setting.

DETAILED DESCRIPTION:
British Columbia is a province which contains four metropolitan areas, each of which contains at least one tertiary care centre that provides Extracorporeal Membrane Oxygenation (ECMO) and cardiovascular surgery services, in addition to critical cardiology services and a coronary catheterization laboratory. Pre-hospital medical care in all areas is provided by British Columbia Emergency Health Services (BCEHS), which uses a tiered system of basic life support and advanced life support (ALS) paramedics (90% of cases have ALS involvement) in coordination with fire department first responders. Medical providers in the study footprint have extensive experience with interventional trials enrolling patients with out-of-hospital cardiac arrest, through participation in the Resuscitation Outcomes Consortium.

Through collaboration of clinicians from all areas and with BCEHS, this study will examine the benefit of a regional ECPR protocol established in one of the metropolitan areas (the "ECPR Protocol Region"), in comparison to the other areas (the "Usual Care Region"). The primary aim is to determine the benefit of incorporating ECPR services into a regional medical system of care for out-of-hospital cardiac arrest. All patients with out-of-hospital cardiac arrest treated by emergency medical services (EMS) in both regions will be prospectively evaluated for study eligibility.

Secondary aims include:

1. To evaluate the effectiveness of ECPR therapy for those with refractory cardiac arrest after 45 minutes of attempted resuscitation.
2. To evaluate the effectiveness of a regional ECPR protocol, in comparison to historical controls.
3. To evaluate the long-term (5-year) outcomes of patients treated with ECPR.
4. To evaluate the quantity of successful organ procurement from those treated with ECPR.
5. To evaluate the cost-effectiveness of a regional ECPR protocol.

This study is a parallel group design with group allocation based on region of treatment. The investigators will compare the outcomes of ECPR-eligible patients in the intervention region, in comparison to patients meeting the same criteria in a comparable setting (the control regions group). Medical care in the control regions will be unaltered by this study.

Group outcomes will be compared. The association of treatment group and outcomes will also be assessed using a logistic regression analysis, while adjusting for other important prognosticators in out-of-hospital cardiac arrest (including initial cardiac rhythm, time to emergency medical services [EMS] arrival, bystander cardiopulmonary resuscitation [CPR], EMS-witnessed arrest, and age).

ELIGIBILITY:
The study evaluates the outcomes of those treated with an ECPR protocol, in comparison to patients in the control region meeting the same criteria. The following is the regional ECPR eligibility criteria:

Inclusion Criteria:

1. Intra-arrest treatment by an ALS paramedic
2. Age ≥ 18 and ≤ 65 years
3. Witnessed arrest
4. Bystander CPR required if initial rhythm is pulseless electrical activity (added to the protocol June, 2018 and applied retrospectively)
5. Cause of the arrest is presumed to be one of the following:

   * No obvious non-cardiac cause is identified
   * Known overdose of one of the following drugs: beta-blocker, calcium channel blocker, tricyclic antidepressants or other psychiatric medications, or digoxin
   * Hypothermia (with T < 32°C)

(5) The patient remains pulseless after a minimum of 3 cycles of CPR (by any professional provider).

Exclusion Criteria:

1. An alternate cause of the arrest is most likely
2. Do Not Resuscitate status
3. Co-morbidities including congestive heart failure, chronic obstructive pulmonary disease or other significant lung disease, dialysis, liver failure (if co-morbidities are unknown to paramedics they will be assumed not present)
4. Active malignancy
5. Pre-existing major neurological deficit
6. Asystole (added to the protocol June, 2018 and applied retrospectively)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Neurological Status will be assessed at hospital discharge using the Cerebral Performance Category scale | Patients will be followed from the time of cardiac arrest until death or hospital discharge, up to 6 months.
  Cerebral Performance Categories 1 and 2 will be considered favourable outcomes. Adjudication for these outcomes will be assessed with a structured algorithm via chart review blinded to treatment group.

SECONDARY OUTCOMES:
Survival will be assessed at hospital discharge | Patients will be followed from the time of cardiac arrest until death or hospital discharge, up to 6 months.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Control Region (Kelowna, Victoria, Fraser Valley), Kelowna, British Columbia
  - BC Emergency Health Services, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No